CLINICAL TRIAL: NCT03454893
Title: An Open-Label, Multinational Study Of The Efficacy And Safety of Ex Vivo, Lentiviral Vector-Mediated Gene Therapy AVR-RD-01 For Treatment-Naive Subjects With Classic Fabry Disease
Brief Title: Open Label, Study Of Efficacy and Safety Of AVR-RD-01 for Treatment-Naive Subjects With Classic Fabry Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: AVROBIO has deprioritized its Fabry disease program
Sponsor: AVROBIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVRO-RD-01-201
Record Dates: First submitted 2017-12-20; First posted 2018-03-06 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Cell therapy; Gene therapy; Lysosomal storage disorder; Lenti-viral
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Assignment AVR-RD-01 (Experimental): AVR-RD-01 is an autologous CD34+-enriched cell fraction transduced with LV/AGA containing an RNA transcript that, after reverse transcription, results in codon-optimized cDNA that, upon its integration into the human genome, encodes for functional human AGA.
  Interventions: Drug: AVR-RD-01

INTERVENTIONS:
Drug: AVR-RD-01 — Single IV infusion of between 3 - 20 x 10^6 CD34+ cells/kg.

SUMMARY:
This was a multinational, open-label study to assess the efficacy and safety of AVR-RD-01 in approximately 15 male subjects, who were 16 years of age or older and postpubertal with a confirmed diagnosis of classic Fabry disease based on deficient alpha galactosidase A (AGA) enzyme activity who were considered treatment naïve, i.e., had not previously received treatment with enzyme replacement therapy (ERT) and/or chaperone therapy within 3 years of the time of Screening.

DETAILED DESCRIPTION:
The duration of each subject's participation in this study was approximately 64 weeks (or 1 year, 12 weeks), comprised of five study periods (Screening, Baseline, Pre-transplant, Transplant, and Post-transplant Follow-up). During the Screening Period (approximately 8 weeks), written informed consent (and assent, if applicable) was obtained and the subject had completed other Screening procedures to confirm study eligibility. Once study eligibility was confirmed, the subjects entered the Baseline Period (up to 3 days) during which time assessments would have been performed to establish a pre-transplant baseline. Once baseline assessments were completed, the subject entered the Pre-transplant Period (approximately 6 weeks) during which time mobilization, apheresis, AVR-RD-01 investigational drug product preparation and testing for release, and conditioning regimen administration to achieve myeloablation took place. Following completion of the Pre-transplant Period, the subject entered the Transplant Period (1 day) during which time AVR-RD-01 infusion took place. After AVR-RD-01 infusion, the subject entered the Post-transplant Follow-up Period (approximately 48 weeks), during which time periodic safety and efficacy assessments were performed to assess measures of engraftment, clinical response, and safety post-transplant.

In January 2022, the study was terminated early due to a decision by the study sponsor, to deprioritize its Fabry disease development program, and therefore, some subjects (n=5) did not complete the study (i.e., Week 48). Subsequently, in August 2023, the long-term follow-up study (AVRO-RD-01-LTF01), was also terminated early due to the decision by the sponsor to terminate the development program for Fabry disease, and therefore, no subjects completed the 15-year long-term follow-up study. This decision to terminate was not based on any safety or medical reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was male, 16 years of age or older (18 years of age or older in the US), and post pubertal,(minimum age by region)
2. Subject had a confirmed diagnosis of classic Fabry disease based on deficient AGA enzyme activity (defined as < 1% of normal).

Exclusion Criteria:

1. Subject had a galactosidase alpha (GLA) gene mutation associated with late-onset cardiac variant Fabry disease.
2. Subject had previously received ERT and/or chaperone therapy within 3 years for treatment of Fabry disease.
3. Subject had tested positive for anti-AGA antibodies at the time of screening.
4. Subject had eGFR < 60 mL/min/1.73 m² (ie, chronic kidney disease [CKD] stage ≥ 3) at Screening.
5. Subject had a prior history of myocardial infarction (MI).
6. Subject had a history of coronary artery disease (CAD) with angina requiring percutaneous transluminal coronary angioplasty (with or without stent placement) and/or coronary artery bypass graft (CABG).
7. Subject had a history of moderate to severe valvular heart disease requiring valve replacement.
8. Subject had a history of heart failure, moderate to severe diastolic dysfunction, and/or left ventricular ejection fraction (LVEF) ≤ 45% on echocardiogram (ECHO) performed at rest at Screening.
9. Subject had a history of clinically significant cardiac arrhythmia (eg, heart block [second or third degree], atrial fibrillation requiring therapy, ventricular fibrillation, ventricular tachycardia, supraventricular tachycardia, or cardiac arrest).

   Note [history of intermittent atrial fibrillation not requiring treatment was allowed].
10. Subject had a prior history of stroke and/or transient ischemic attack (TIA).
11. Subject had aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal (ULN) at Screening.
12. Subject had a prior history of (or current) malignancy; the one exception is a prior history of resected basal cell carcinoma.
13. Subject had previously received treatment with AVR-RD-01 or any other gene therapy.

Other inclusion/exclusion criteria apply.

Ages: 16 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inderpal Panesar, MRPharmS, Study Director — AVROBIO, Inc
Locations (5):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Royal Melbourne Hospital, Melbourne, Parkville VIC
  - Royal Perth Hospital, Perth
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of subjects who signed the ICF was 16 (one subject who re-screened was not considered enrolled initially), as a result there were 15 distinct subjects who signed ICF. There were 4 participants who failed screening and were not rescreened.
  The Safety population consists of all 11 enrolled subjects who received any preparatory medication.
  The Infused population consists of all 9 enrolled subjects who received all preparatory medications and AVR-RD-01.
Groups:
- Single Assignment AVR-RD-01: AVR-RD-01 is an autologous CD34+-enriched cell fraction transduced with LV/AGA containing an RNA transcript that, after reverse transcription, results in codon-optimized cDNA that, upon its integration into the human genome, encodes for functional human AGA.
  Drug: AVR-RD-01 Single IV infusion of between 3 - 20 x 10^6 CD34+ cells/kg
Period: Overall Study
Arm/Group | Single Assignment AVR-RD-01
Started | 15
Safety Population | 11
Infused Population | 9
Completed | 6
Not Completed | 9
Not completed — Study Terminated by the Sponsor | 5
Not completed — Did not pass screening | 4

BASELINE CHARACTERISTICS:
Population: Safety population consists of all enrolled subjects who received any preparatory medication.
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.45 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The AE/SAE are also inclusive of any abnormalities in Clinical Laboratory Tests, Vital Signs and in Electrocardiographs (ECGs). Of the 13 serious adverse events, no SAEs reported were considered related to AVR RD 01. Of the 354 adverse events, no AEs were considered related to AVR RD 01. The SAEs and AEs reported in the study were attributed to the conditioning agent used, the underlying disease, comorbid conditions, study procedures and concomitant medications.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Safety population consists of all enrolled subjects who received any preparatory medication.
Measure: Number; unit: Number of events
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 11
Number of events
  AE | 354
  SAE | 13

2. Primary Outcome: Change From Baseline in Immunogenicity of AVR-RD-01
Description: Number of subjects with changes in anti-AGA antibodies from Baseline to post infusion timepoints. Unite of measure: Number of subjects negative at baseline but positive at post-treatment timepoints. A negative or zero result (titer lower or unchanged at post-infusion timepoints compare to Baseline) indicates no immune response to the therapeutic protein.
Time Frame: Baseline to Week 48 post gene therapy
Population: The infused population includes all enrolled subjects who received preparatory medications and AVR-RD-01. Four tested positive for anti-AGA antibodies post-AVR-RD-01 infusion at Week 48 or Early Termination visit.
Measure: Number; unit: Number of positive subjects
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
Number of positive subjects | 4

3. Primary Outcome: Presence of Replication Competent Lentivirus (RCL)
Description: The "Presence of RCL" is a theoretical risk of lentiviral gene therapy treatment based on the theory that it may be possible for inadvertent generation of RCL caused either by recombination of the lentiviral vector plasmids during the vector production process or by mobilization of proviral DNA in vivo by infectious retroviruses (HIV). The absence of RCL is a positive indicator of safety.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Number; unit: Number of positive subjects
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
Number of positive subjects | 0

4. Primary Outcome: Evaluation of Aberrant Clonal Expansion
Description: Integration Site Analysis (ISA) uses next generation sequencing to identify junction sites between the integrated therapeutic transgene and the host genome. Samples are analyzed for the emergence of clonality (defined as (a single clone accounting for greater than 20% of the population) and whether any integration site is within or near a known oncogene.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Number; unit: number of abnormal clonal proliferations
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
number of abnormal clonal proliferations | 0

5. Primary Outcome: Change From Baseline in the Average Number of Gb3 Inclusions (ie, Myelinosomes) Per Kidney Peritubular Capillary (PTC) Per Subject
Description: Globotriaosylceramide (Gb3) Inclusions in Peritubular Capillaries (PTC) on Kidney Biopsy. Electron microscopic images of kidney biopsy samples were taken and read centrally by two independent renal pathologists, each of whom scored the average number of Gb3 inclusions per kidney PTC per subject using a quantification method. Healthy renal tissue would have no Gb3 inclusions. A reduction from baseline is desirable.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01. Of the nine subjects, only 2 subjects had baseline and Week 48 results to measure change from baseline. The remaining seven subjects either did not provide both samples or the samples provided were not evaluable.
Measure: Mean (Full Range); unit: Number of inclusions
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 2
Number of inclusions | -3.555 [-4.020 to -3.090]

6. Secondary Outcome: Average Vector Copy Number (VCN) in Peripheral Blood Leukocytes as Assessed by Quantitative Polymerase Chain Reaction (qPCR) and/or Droplet Digital Polymerase Chain Reaction (ddPCR)
Description: Vector Copy Number (VCN) is a measurement of the number of copies of the therapeutic transgene found in a sample, relative to copies of a reference gene in the human genome. This is an estimate of the number of integration sites per cell (on average). A VCN of 1 would signify that a sample of cells evaluated contains on average at least one [working] copy of the therapeutic transgene per cell.
Time Frame: At Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: copies/diploid genome
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
copies/diploid genome
  Week 24: number analyzed (Participants) | 8
  Week 24 | 0.383 (0.4628)
  Week 48: number analyzed (Participants) | 7
  Week 48 | 0.313 (0.3447)

7. Secondary Outcome: Change From Baseline (CFB) in AGA Enzyme Activity Level in Plasma and Peripheral Blood Leukocytes (PBLs)
Description: Treatment-naïve Fabry patients are deficient in alpha-galactosidase A (AGA) enzyme activity due to mutations in the GLA gene. Any therapeutic option offered should aim to increase the amount of available AGA enzyme. This assay measured the AGA enzyme activity levels in plasma and PBLs. It should be noted that the measurement in plasma reflects the amount of "free" AGA enzyme that has been released from cells into the extracellular space and is therefore considered a more indirect measure of AGA enzyme activity, compared to the result in PBLs which is more of a direct measure of enzyme within cells. In both cases, enzyme activity is expected to increase from Baseline to the post-infusion timepoints.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: nmol/h/mg
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
nmol/h/mg
  CFB Plasma W24: number analyzed (Participants) | 7
  CFB Plasma W24 | 1.973 (2.585)
  CFB Plasma W48: number analyzed (Participants) | 6
  CFB Plasma W48 | 1.548 (2.152)
  CFB PBL Week 24: number analyzed (Participants) | 8
  CFB PBL Week 24 | 29.524 (39.194)
  CFB PBL Week 48: number analyzed (Participants) | 7
  CFB PBL Week 48 | 18.973 (32.800)

8. Secondary Outcome: Change From Baseline in Globotriaosylceramide (Gb3) Biomarkers for Fabry Disease in Plasma
Description: Globotriaosylceramide (Gb3) is the substrate that accumulates in the lysosomes of patients affected by Fabry Disease as a result of deficiencies in AGA enzyme activity. Treatment-naive patients are expected to have high levels of Gb3 in their lysosomes and correspondingly elevated levels in plasma. Treatment with AVR-RD-01 is intended to replace the missing AGA enzymatic activity, which allows degradation of accumulated Gb3 substrate in the lysosomes and reductions in the levels of circulating Gb3 in plasma.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
nM
  Week 24: number analyzed (Participants) | 8
  Week 24 | -3334.0 (3846.8)
  Week 48: number analyzed (Participants) | 5
  Week 48 | -5067.8 (4067.0)

9. Secondary Outcome: Change From Baseline in Globotriaosylceramide (Gb3) Biomarkers for Fabry Disease in Urine
Description: Globotriaosylceramide (Gb3) is the substrate that accumulates in the lysosomes of patients affected by Fabry Disease as a result of deficiencies in AGA enzyme activity. Treatment-naive patients are expected to have high levels of Gb3 in their lysosomes and correspondingly elevated levels in urine. Treatment with AVR-RD-01 is intended to replace the missing AGA enzymatic activity, which allows degradation of accumulated Gb3 substrate in the lysosomes and reductions in the levels of excreted Gb3 in urine.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: nmol/mmol creatinine
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
nmol/mmol creatinine
  Week 24 | -11.73 (309.78)
  Week 48 | -188.73 (262.90)

10. Secondary Outcome: Change From Baseline in Substrate (i.e. Gb3) in Skin Biopsy
Description: Globotriaosylceramide (Gb3) is the substrate that accumulates in the lysosomes of patients affected by Fabry Disease as a result of deficiencies in AGA enzyme activity. Treatment-naive patients are expected to have high levels of Gb3 in their lysosomes and correspondingly elevated levels in tissue samples. Treatment with AVR-RD-01 is intended to replace the missing AGA enzymatic activity, which allows degradation of accumulated Gb3 substrate in the lysosomes and reductions in the levels of measured Gb3 in tissues.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: number of myelinosomes
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
number of myelinosomes
  Myelinosomes in superficial dermal capillary endothelial cells (Week 24) | -0.4 (1.3)
  Myelinosomes in superficial dermal capillary endothelial cells (Week 48) | -0.5 (1.0)
  Myelinosomes in deep dermal capillary endothelial cells (Week 24) | 0 (1.3)
  Myelinosomes in deep dermal capillary endothelial cells (Week 48) | -0.5 (1.0)
  Myelinosomes in vascular smooth muscle cells (Week 24) | 0.1 (1.2)
  Myelinosomes in vascular smooth muscle cells (Week 48) | -0.5 (1.0)
  Myelinosomes in perineurium (Week 24) | 0 (1.4)
  Myelinosomes in perineurium (Week 48) | -0.5 (1.0)

11. Secondary Outcome: Change From Baseline in Renal Function as Assessed by Measured Glomerular Filtration Rate (mGFR)
Description: mGFR is a measure of the time the kidney takes to filter products that the body does not naturally produce.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
mL/min/1.73m^2 | -2.358 (14.502)

12. Secondary Outcome: Change From Baseline in Renal Function as Assessed by Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR is the measure to evaluate kidney function. It is the estimated amount of blood that is filtered through all glomeruli in a given time.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
mL/min/1.73 m^2
  Week 24 | -6.386 (9.699)
  Week 48 | -3.561 (7.332)

13. Secondary Outcome: Change From Baseline in Renal Function as Assessed by Urine Total Protein Levels
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01. No data were collected for any subjects since samples were not analyzed in order to produce data (Refer to "Limitations and Caveat" section.")
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline in Renal Function as Assessed by Urine Albumin Levels
Description: A healthy kidney only allows very small amounts of albumin to pass from the blood into the urine. An increased level of albumin in urine (albuminuria) is a marker of renal damage.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
mg/dL
  Week 24 | 0.915 (6.704)
  Week 48 | 0.643 (5.789)

15. Secondary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) as Assessed by Cardiac Magnetic Resonance Imaging (MRI)
Description: LVMI is a surrogate of left ventricular hypertrophy. An increase in LVMI is an independent risk factor for cardiovascular morbidity and mortality.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
g/m^2 | 7.270 (6.055)

16. Secondary Outcome: Change From Baseline in Abdominal Pain and Stool Consistency as Assessed by the Diary for Irritable Bowel Syndrome Symptoms-Diarrhea (DIBSS-D)
Description: DIBSS-D assesses bowel habits and abdominal symptoms over a period of time. It was administered daily for 14 days commencing at each study visit.
  Stool Consistency scale has been converted to a numeric rating scale for ease of analysis, where 1=Very hard; 2=Hard; 3=Neither too hard nor too soft; 4=Loose but not lumpy; 5=Very loose and watery. The median of each 14-day period was derived per patient, per visit before deriving the group median. Group median at Baseline (pre-treatment) was 3.540 (n=9). Change from baseline (CFB) is presented below. An increase CFB indicates softening of the stools, and a decrease CFB indicates hardening of the stools. Abdominal Pain measure asked the patient to rate the worst level of pain within the past 24hrs (0=no pain; 10=worst possible pain). A mean score was derived for each 14-day period per patient, per visit, and these means used to derive a group mean. An increase CFB indicates more abdominal pain; a decrease CFB indicates less abdominal pain.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
units on a scale
  Abdominal Pain Week 24 | -0.445 (0.583)
  Abdominal Pain Week 48 | -0.497 (0.626)
  Stool Consistency Week 24 | -0.373 (0.216)
  Stool Consistency Week 48 | -0.530 (0.104)

17. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-SF) Questionnaire Scores
Description: The short version of the BPI (Short form) includes 9 items: Q1 - Q9, Question 9 includes 7 sub-items (Q9a - Q9g). It uses a 0 to 10 numeric rating scales for item rating. The pain severity score is calculated as the average of questions answered: Q3 (worst pain), Q4 (least pain), Q5 (average pain) and Q6 (current pain). The pain interference score is calculated as the average of the answered Q9 sub-items, which represents pain interference with general activity (Q9a), mood (Q9b), walking ability (Q9c), normal work (Q9d), relations with other people (Q9e), sleep (Q9f), and enjoyment of life (Q9g). A reduction in score from baseline indicates less pain.
Time Frame: Baseline to Week 24 and Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
score on a scale
  Week 24 (pain severity): number analyzed (Participants) | 8
  Week 24 (pain severity) | -0.188 (0.874)
  Week 48 (pain severity): number analyzed (Participants) | 6
  Week 48 (pain severity) | -0.500 (0.612)
  Week 24 (pain interference): number analyzed (Participants) | 6
  Week 24 (pain interference) | 0.073 (1.007)
  Week 48 (pain interference): number analyzed (Participants) | 6
  Week 48 (pain interference) | -0.573 (0.996)

18. Secondary Outcome: Change From Baseline in Physical and Mental Functioning as Assessed by the Short Form 36 (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The original version of the SF-36 was administered to the participants and consisted of eight subscales (Vitality, Physical Functioning, Bodily Pain, General Health Perceptions, Physical Role Functioning, Emotional Role Functioning, Social Role Functioning and Mental Health) each scored from 0 (worst health) to 100 (best heath). These scores were normalized (re-scaled) against mean scores obtained in the US general population (Mean=50, Standard deviation 10). The summary health components PCS and MCS are derived from the eight subscales mentioned above and summarize information from all eight subscales but with different weights. For PCS, highest weights are given to the physical subscales while some mental subscales are given negative weights. For MCS, highest weights are given to the mental subscales while some physical subscales are given negative weights. An increase in the normalized score from baseline indicates improvement in physical and mental functioning.
Time Frame: Baseline to Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01. For Week 24 data, please see comment in "Limitations and Caveats" section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 9
score on a scale
  Physical Functioning Week 48 | 3.235 (4.810)
  Mental Functioning Week 48 | -1.580 (4.652)

19. Secondary Outcome: Average Vector Copy Number (VCN) in Bone Marrow / Progenitor Cells as Assessed by Quantitative Polymerase Chain Reaction (qPCR) and/or Droplet Digital Polymerase Chain Reaction (ddPCR)
Description: VCN is defined as the average number of copies of the therapeutic gene (transgene) in a sample of cells and is a measurement of the number of copies of the vector found in a sample, relative to copies of a reference gene in the human genome. This is an estimate of the number of integration sites per cell (on average). A VCN of 1 would signify that a sample of cells evaluated contains on average at least one [working] copy of the therapeutic transgene per cell. This measurement was for VCN in a sample of Bone marrow progenitor cells obtained from an aspirate.
Time Frame: At Week 48 post gene therapy
Population: The Infused population consists of all enrolled subjects who received all preparatory medications and AVR-RD-01. No analysis performed (refer to "Limitations and Caveats" section)
Measure: Mean (Full Range); unit: copies/diploid genome
Arm/Group | Single Assignment AVR-RD-01
Number analyzed (Participants) | 1
copies/diploid genome | 1.14 [1.14 to 1.14]

ADVERSE EVENTS:
Time Frame: Up to week 48
Description: Of the 13 serious adverse events, no SAEs reported were considered related to AVR RD 01. Of the 354 adverse events, no AEs were considered related to AVR RD 01. The SAEs and AEs reported in the study were attributed to the conditioning agent used, the underlying disease, comorbid conditions, study procedures and concomitant medications.
Groups:
- Single Assignment AVR-RD-01: AVR-RD-01 is an autologous CD34+-enriched cell fraction transduced with LV/AGA containing an RNA transcript that, after reverse transcription, results in codon-optimized cDNA that, upon its integration into the human genome, encodes for functional human.
  Drug: AVR-RD-01 Single IV infusion of between 3 - 20 x 10^6 CD34+ cells/kg.
Arm/Group | Single Assignment AVR-RD-01
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Assignment AVR-RD-01 (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Assignment AVR-RD-01 (N=11)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 9 (11)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 9 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Fabry's disease (Congenital, familial and genetic disorders) | 1 (2)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Primary hypogonadism (Endocrine disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6)
Dental caries (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (15)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (10)
Face oedema (General disorders) | 1 (2)
Fatigue (General disorders) | 2 (2)
Feeling abnormal (General disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (3)
Injection site induration (General disorders) | 1 (3)
Injection site pain (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 5 (5)
Nodule (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 5 (6)
Vaccination site pain (General disorders) | 2 (3)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Immunisation reaction (Immune system disorders) | 1 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2)
Gingivitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1)
Citrate toxicity (Injury, poisoning and procedural complications) | 6 (7)
Meniscus cyst (Injury, poisoning and procedural complications) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (9)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site erythema (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site pain (Injury, poisoning and procedural complications) | 4 (5)
Alanine aminotransferase increased (Investigations) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (5)
Blood follicle stimulating hormone increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 2 (2)
Cardiac murmur (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
Urine analysis abnormal (Investigations) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 (4)
Abnormal weight gain (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (9)
Lethargy (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Depressed mood (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Azoospermia (Reproductive system and breast disorders) | 5 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Oligospermia (Reproductive system and breast disorders) | 1 (1)
Scrotal discomfort (Reproductive system and breast disorders) | 1 (1)
Scrotal erythema (Reproductive system and breast disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
SF-36 data at W24 was inadvertently not collected due to omission in the Protocol Schedule of Assessments.

Invasive sampling, such as bone marrow aspirate, was only provided by one subject at Week 48.

Central laboratory only reported albumin levels in urine and not urine total protein data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03454893/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03454893/SAP_003.pdf